CLINICAL TRIAL: NCT02121496
Title: Social Circumstances, Parenting Techniques, and Infant Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: The Robin Hood Foundation (Unknown)
Responsible Party: Principal Investigator, Catherine Monk, Professor of Medical Psychology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #6889
Record Dates: First submitted 2014-03-28; First posted 2014-04-23 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Postpartum Depression; Infant Development; Rhythm; Sleep
Keywords: Depression; Development; Infant sleep
MeSH Terms: conditions — Depression, Postpartum; Depression | interventions — Health Resources

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resources for Postpartum Parenting (Experimental): Behavioral intervention will include techniques to help mothers get their infants to cry/fuss less and sleep more to determine if this has an effect on prevalence of postpartum depression in low SES women and if it improves the quality of mother-infant interaction and subsequent child development.
  Interventions: Behavioral: Resources for Postpartum Parenting
- Control Group (No Intervention): This group will not receive the coaching tips to help babies cry less and sleep more.

INTERVENTIONS:
Behavioral: Resources for Postpartum Parenting — The intervention includes four-sessions that targets maternal caregiving of young infants to increase infant sleep and reduce fuss/cry behavior and thereby simultaneously consolidate women's enjoyment of and confidence in their maternal role, this, in turn, promotes a cycle of a mutually re- warding engagement in the mother-infant dyad - the antithesis of a 'toxic' experience, and a strong foundation for improving the chances of a successful psychosocial adjustment, including adequate employment. Investigators believe PREPP holds tremendous promise as an intervention to fill the science-practice gap in the promotion of an optimal emotional environment for the developing infant, particularly for women and children living in poverty and/or facing significant psychosocial hardship.
  Other Names: Practical Resources for Effective Postpartum Parenting
  Arms: Resources for Postpartum Parenting

SUMMARY:
1. Investigators aim to assess a novel behavioral intervention (currently approved in Protocol #6285) behavioral intervention that promotes maternally-mediated behavioral changes in young infants to reduce the risk of postpartum depression in a group of low income women. More specifically, investigators aim to determine if a behavioral intervention targeting maternal caregiving of young infants can increase infant sleep and reduce fuss/cry behavior and thereby: (1) reduce the incidence and/or severity of postpartum maternal depression in low socioeconomic status (SES) women, and (2) improve the quality of mother-infant interaction and subsequent child development. Investigators will study:

   1. The feasibility of applying this protocol with a low SES population
   2. The effectiveness of the intervention compared to usual care
   3. If the effects of the intervention can be detected in assessments of the quality of mother-infant interaction and infant neurocognitive development
2. Investigators aim to determine whether this behavioral intervention can affect infant development as measured by neurodevelopmental assessments and cortisol reactivity at 4 months of age.

DETAILED DESCRIPTION:
Developmental research consistently shows that postpartum depression has a negative impact on cognitive and emotional development during infancy and childhood. Low SES women face unique stressors and social challenges. Rates of postpartum depression are significantly higher in this group (23-33%) than in the general population (10-15%).

The purpose of this study is to understand how social circumstances, women's mood, and parenting techniques affect infant and child development. Specifically, investigators are interested in finding out whether a behavioral intervention, already being administered in IRB approved protocol #6285, targeting maternal caregiving of young infants can increase infant sleep and reduce fuss/cry behavior, thereby reducing the incidence and/or severity of maternal depression and anxiety symptoms, improving the quality of the mother-infant interaction, and improving infant developmental outcomes.

By collecting stress reports from women from low SES backgrounds during pregnancy and the postpartum period and by conducting follow-up observational assessments of the quality of mother-infant interaction, infant learning, infant cortisol reactivity, and infant neurocognitive development, investigators hope to identify whether this intervention can effectively meet these aims.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women between 24 and 38 weeks gestation (based on self-report)
* Ages 18-45 (based on self-report) 3. English speaking (based on self-report)
* Salary indicated to be at New York City standardized "Struggling level" or lower - $47,700 annual for a family of 4 (based on self-report)
* Experiencing one or more of nine social adversity hardships (based on self report)
* Experiencing a healthy pregnancy, free from any significant medical complication (based on self-report)
* Receiving standard prenatal care (based on self-report)

Exclusion Criteria:

* Multi-fetal pregnancy (based on self-report)
* Smoking, illicit drug use, or alcohol use during pregnancy (based on self-report)
* Acute medical illness or significant pregnancy complication (based on self-report)
* Currently in weekly, individual psychotherapy - group therapy and psychiatric management ok (based on self-report)
* Psychotic d/o; Bipolar I; Major Depressive d/o (based on M.I.N.I.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in maternal mood and prevalence/severity of postpartum depression. | 6 weeks postpartum, 10 weeks postpartum, 16 weeks postpartum
  Investigators will be assessing and tracking the incidence and/or severity of postpartum depression with the use of mood and stress questionnaires (Hamilton Depression Scale, Hamilton Anxiety Scale, Perceived Stress Scale, Center for Epidemiological Studies Depression Scale) administered at 4-6 weeks postpartum, 10 weeks postpartum, and 16 weeks postpartum.

SECONDARY OUTCOMES:
The effect of behavioral intervention for infants on infant development | 4 months (infant age)
  Investigators will use neurodevelopmental assessments (Bayley Scale of Infant Development, Still Face Protocol, Free Play Observation, and Conjugate Kicking Task) and cortisol reactivity to assess infant development at 4 months of age.
The effect of behavioral intervention on infant sleep and fuss behavior | 6 weeks, 4 months (infant age)
  The infant's sleep and fuss/cry behavior will be assessed at 6 weeks and 16 weeks of age (Baby Day Diary)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Monk, Ph.D., Principal Investigator — NYPI, CUMC
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Peng, S. S. High School Dropouts: A National Concern. (National Center for Education Statistics, Washington, D.C., 1985).
- [Background] Markham JA, Greenough WT. Experience-driven brain plasticity: beyond the synapse. Neuron Glia Biol. 2004 Nov;1(4):351-63. doi: 10.1017/s1740925x05000219. PMID 16921405
- [Background] Nelson CA, Bloom FE. Child Development and Neuroscience. Child Dev. 1997 Oct;68(5):970-987. doi: 10.1111/j.1467-8624.1997.tb01974.x. PMID 29106726
- [Background] Whiffen VE, Gotlib IH. Infants of postpartum depressed mothers: temperament and cognitive status. J Abnorm Psychol. 1989 Aug;98(3):274-9. doi: 10.1037//0021-843x.98.3.274. PMID 2768663
- [Background] Doan SN, Evans GW. Maternal responsiveness moderates the relationship between allostatic load and working memory. Dev Psychopathol. 2011 Aug;23(3):873-80. doi: 10.1017/S0954579411000368. PMID 21756438
- [Background] Shonkoff JP, Garner AS; Committee on Psychosocial Aspects of Child and Family Health; Committee on Early Childhood, Adoption, and Dependent Care; Section on Developmental and Behavioral Pediatrics. The lifelong effects of early childhood adversity and toxic stress. Pediatrics. 2012 Jan;129(1):e232-46. doi: 10.1542/peds.2011-2663. Epub 2011 Dec 26. PMID 22201156
- [Background] Garner AS, Shonkoff JP; Committee on Psychosocial Aspects of Child and Family Health; Committee on Early Childhood, Adoption, and Dependent Care; Section on Developmental and Behavioral Pediatrics. Early childhood adversity, toxic stress, and the role of the pediatrician: translating developmental science into lifelong health. Pediatrics. 2012 Jan;129(1):e224-31. doi: 10.1542/peds.2011-2662. Epub 2011 Dec 26. PMID 22201148
- [Background] Tau GZ, Peterson BS. Normal development of brain circuits. Neuropsychopharmacology. 2010 Jan;35(1):147-68. doi: 10.1038/npp.2009.115. PMID 19794405
- [Background] Vaughn B, Egeland B, Sroufe LA, Waters E. Individual differences in infant-mother attachment at twelve and eighteen months: stability and change in families under stress. Child Dev. 1979 Dec;50(4):971-5. PMID 535447
- [Background] Sroufe LA. Psychopathology as an outcome of development. Dev Psychopathol. 1997 Spring;9(2):251-68. doi: 10.1017/s0954579497002046. PMID 9201444
- [Background] Sroufe LA. Attachment and development: a prospective, longitudinal study from birth to adulthood. Attach Hum Dev. 2005 Dec;7(4):349-67. doi: 10.1080/14616730500365928. PMID 16332580
- [Background] Meaney MJ, Diorio J, Francis D, Widdowson J, LaPlante P, Caldji C, Sharma S, Seckl JR, Plotsky PM. Early environmental regulation of forebrain glucocorticoid receptor gene expression: implications for adrenocortical responses to stress. Dev Neurosci. 1996;18(1-2):49-72. doi: 10.1159/000111395. PMID 8840086
- [Background] Meaney MJ, Szyf M, Seckl JR. Epigenetic mechanisms of perinatal programming of hypothalamic-pituitary-adrenal function and health. Trends Mol Med. 2007 Jul;13(7):269-77. doi: 10.1016/j.molmed.2007.05.003. Epub 2007 Jun 4. PMID 17544850
- [Background] Szyf M, Weaver I, Meaney M. Maternal care, the epigenome and phenotypic differences in behavior. Reprod Toxicol. 2007 Jul;24(1):9-19. doi: 10.1016/j.reprotox.2007.05.001. Epub 2007 May 10. PMID 17561370
- [Background] Grossman AW, Churchill JD, McKinney BC, Kodish IM, Otte SL, Greenough WT. Experience effects on brain development: possible contributions to psychopathology. J Child Psychol Psychiatry. 2003 Jan;44(1):33-63. doi: 10.1111/1469-7610.t01-1-00102. PMID 12553412
- [Background] Francis D, Diorio J, Liu D, Meaney MJ. Nongenomic transmission across generations of maternal behavior and stress responses in the rat. Science. 1999 Nov 5;286(5442):1155-8. doi: 10.1126/science.286.5442.1155. PMID 10550053
- [Background] Caldji C, Diorio J, Meaney MJ. Variations in maternal care in infancy regulate the development of stress reactivity. Biol Psychiatry. 2000 Dec 15;48(12):1164-74. doi: 10.1016/s0006-3223(00)01084-2. PMID 11137058
- [Background] Lupien SJ, McEwen BS, Gunnar MR, Heim C. Effects of stress throughout the lifespan on the brain, behaviour and cognition. Nat Rev Neurosci. 2009 Jun;10(6):434-45. doi: 10.1038/nrn2639. Epub 2009 Apr 29. PMID 19401723
- [Background] McEwen BS. Steroid hormones: effect on brain development and function. Horm Res. 1992;37 Suppl 3:1-10. doi: 10.1159/000182393. PMID 1330863
- [Background] Ouellet-Morin I, Boivin M, Dionne G, Lupien SJ, Arseneault L, Barr RG, Perusse D, Tremblay RE. Variations in heritability of cortisol reactivity to stress as a function of early familial adversity among 19-month-old twins. Arch Gen Psychiatry. 2008 Feb;65(2):211-8. doi: 10.1001/archgenpsychiatry.2007.27. PMID 18250259
- [Background] Evans GW, Gonnella C, Marcynyszyn LA, Gentile L, Salpekar N. The role of chaos in poverty and children's socioemotional adjustment. Psychol Sci. 2005 Jul;16(7):560-5. doi: 10.1111/j.0956-7976.2005.01575.x. PMID 16008790
- [Background] Brennan PA, Le Brocque R, Hammen C. Maternal depression, parent-child relationships, and resilient outcomes in adolescence. J Am Acad Child Adolesc Psychiatry. 2003 Dec;42(12):1469-77. doi: 10.1097/00004583-200312000-00014. PMID 14627882
- [Background] Bradley RH, Whiteside L, Mundfrom DJ, Casey PH, Kelleher KJ, Pope SK. Early indications of resilience and their relation to experiences in the home environments of low birthweight, premature children living in poverty. Child Dev. 1994 Apr;65(2 Spec No):346-60. PMID 8013226
- [Background] Luthar SS, Cicchetti D, Becker B. The construct of resilience: a critical evaluation and guidelines for future work. Child Dev. 2000 May-Jun;71(3):543-62. doi: 10.1111/1467-8624.00164. PMID 10953923
- [Background] Evans GW, Kim P, Ting AH, Tesher HB, Shannis D. Cumulative risk, maternal responsiveness, and allostatic load among young adolescents. Dev Psychol. 2007 Mar;43(2):341-51. doi: 10.1037/0012-1649.43.2.341. PMID 17352543
- [Background] Kaplan LA, Evans L, Monk C. Effects of mothers' prenatal psychiatric status and postnatal caregiving on infant biobehavioral regulation: can prenatal programming be modified? Early Hum Dev. 2008 Apr;84(4):249-56. doi: 10.1016/j.earlhumdev.2007.06.004. Epub 2007 Aug 30. PMID 17761394
- [Background] Bernier A, Carlson SM, Whipple N. From external regulation to self-regulation: early parenting precursors of young children's executive functioning. Child Dev. 2010 Jan-Feb;81(1):326-39. doi: 10.1111/j.1467-8624.2009.01397.x. PMID 20331670
- [Background] Kochanska G, Murray KT. Mother-child mutually responsive orientation and conscience development: from toddler to early school age. Child Dev. 2000 Mar-Apr;71(2):417-31. doi: 10.1111/1467-8624.00154. PMID 10834474
- [Background] Kochanska G, Coy KC, Murray KT. The development of self-regulation in the first four years of life. Child Dev. 2001 Jul-Aug;72(4):1091-111. doi: 10.1111/1467-8624.00336. PMID 11480936
- [Background] Aksan N, Kochanska G, Ortmann MR. Mutually responsive orientation between parents and their young children: toward methodological advances in the science of relationships. Dev Psychol. 2006 Sep;42(5):833-48. doi: 10.1037/0012-1649.42.5.833. PMID 16953690
- [Background] Kochanska G, Philibert RA, Barry RA. Interplay of genes and early mother-child relationship in the development of self-regulation from toddler to preschool age. J Child Psychol Psychiatry. 2009 Nov;50(11):1331-8. doi: 10.1111/j.1469-7610.2008.02050.x. Epub 2009 Jan 12. PMID 19207629
- [Background] Feldman R. From biological rhythms to social rhythms: Physiological precursors of mother-infant synchrony. Dev Psychol. 2006 Jan;42(1):175-88. doi: 10.1037/0012-1649.42.1.175. PMID 16420127
- [Background] Feldman R. Parent-infant synchrony and the construction of shared timing; physiological precursors, developmental outcomes, and risk conditions. J Child Psychol Psychiatry. 2007 Mar-Apr;48(3-4):329-54. doi: 10.1111/j.1469-7610.2006.01701.x. PMID 17355401
- [Background] Hunziker UA, Barr RG. Increased carrying reduces infant crying: a randomized controlled trial. Pediatrics. 1986 May;77(5):641-8. PMID 3517799
- [Background] Pinilla T, Birch LL. Help me make it through the night: behavioral entrainment of breast-fed infants' sleep patterns. Pediatrics. 1993 Feb;91(2):436-44. PMID 8424024
- [Background] St James-Roberts I, Sleep J, Morris S, Owen C, Gillham P. Use of a behavioural programme in the first 3 months to prevent infant crying and sleeping problems. J Paediatr Child Health. 2001 Jun;37(3):289-97. doi: 10.1046/j.1440-1754.2001.00699.x. PMID 11468047
- [Background] van Sleuwen BE, Engelberts AC, Boere-Boonekamp MM, Kuis W, Schulpen TW, L'Hoir MP. Swaddling: a systematic review. Pediatrics. 2007 Oct;120(4):e1097-106. doi: 10.1542/peds.2006-2083. PMID 17908730
- [Background] Braveman P, Marchi K, Egerter S, Kim S, Metzler M, Stancil T, Libet M. Poverty, near-poverty, and hardship around the time of pregnancy. Matern Child Health J. 2010 Jan;14(1):20-35. doi: 10.1007/s10995-008-0427-0. Epub 2008 Nov 27. PMID 19037715
- [Background] Paybarah, A. in The New York Observer (New York 2008).
- [Background] Werner E, Zhao Y, Evans L, Kinsella M, Kurzius L, Altincatal A, McDonough L, Monk C. Higher maternal prenatal cortisol and younger age predict greater infant reactivity to novelty at 4 months: an observation-based study. Dev Psychobiol. 2013 Nov;55(7):707-18. doi: 10.1002/dev.21066. Epub 2012 Jul 6. PMID 22778036
- [Background] Slade A, Sadler L, De Dios-Kenn C, Webb D, Currier-Ezepchick J, Mayes L. Minding the baby a reflective parenting program. Psychoanal Study Child. 2005;60:74-100. doi: 10.1080/00797308.2005.11800747. PMID 16649676
- [Background] Cassidy J, Ziv Y, Stupica B, Sherman LJ, Butler H, Karfgin A, Cooper G, Hoffman KT, Powell B. Enhancing attachment security in the infants of women in a jail-diversion program. Attach Hum Dev. 2010 Jul;12(4):333-53. doi: 10.1080/14616730903416955. PMID 20582844
- [Background] Olds D, Henderson CR Jr, Cole R, Eckenrode J, Kitzman H, Luckey D, Pettitt L, Sidora K, Morris P, Powers J. Long-term effects of nurse home visitation on children's criminal and antisocial behavior: 15-year follow-up of a randomized controlled trial. JAMA. 1998 Oct 14;280(14):1238-44. doi: 10.1001/jama.280.14.1238. PMID 9786373
- [Background] Olds DL, Sadler L, Kitzman H. Programs for parents of infants and toddlers: recent evidence from randomized trials. J Child Psychol Psychiatry. 2007 Mar-Apr;48(3-4):355-91. doi: 10.1111/j.1469-7610.2006.01702.x. PMID 17355402
- [Background] Olds DL, Eckenrode J, Henderson CR Jr, Kitzman H, Powers J, Cole R, Sidora K, Morris P, Pettitt LM, Luckey D. Long-term effects of home visitation on maternal life course and child abuse and neglect. Fifteen-year follow-up of a randomized trial. JAMA. 1997 Aug 27;278(8):637-43. PMID 9272895
- [Background] Olds DL, Kitzman H, Hanks C, Cole R, Anson E, Sidora-Arcoleo K, Luckey DW, Henderson CR Jr, Holmberg J, Tutt RA, Stevenson AJ, Bondy J. Effects of nurse home visiting on maternal and child functioning: age-9 follow-up of a randomized trial. Pediatrics. 2007 Oct;120(4):e832-45. doi: 10.1542/peds.2006-2111. PMID 17908740
- [Background] Eckenrode J, Campa M, Luckey DW, Henderson CR Jr, Cole R, Kitzman H, Anson E, Sidora-Arcoleo K, Powers J, Olds D. Long-term effects of prenatal and infancy nurse home visitation on the life course of youths: 19-year follow-up of a randomized trial. Arch Pediatr Adolesc Med. 2010 Jan;164(1):9-15. doi: 10.1001/archpediatrics.2009.240. PMID 20048236
- [Background] Miller AR, Barr RG, Eaton WO. Crying and motor behavior of six-week-old infants and postpartum maternal mood. Pediatrics. 1993 Oct;92(4):551-8. PMID 8414826
- [Background] Barr RG, Kramer MS, Boisjoly C, McVey-White L, Pless IB. Parental diary of infant cry and fuss behaviour. Arch Dis Child. 1988 Apr;63(4):380-7. doi: 10.1136/adc.63.4.380. PMID 3365007
- [Background] Kochanska G, Aksan N. Development of mutual responsiveness between parents and their young children. Child Dev. 2004 Nov-Dec;75(6):1657-76. doi: 10.1111/j.1467-8624.2004.00808.x. PMID 15566371
- [Background] Meins E, Fernyhough C, Fradley E, Tuckey M. Rethinking maternal sensitivity: mothers' comments on infants' mental processes predict security of attachment at 12 months. J Child Psychol Psychiatry. 2001 Jul;42(5):637-48. PMID 11464968
- [Background] Biringen Z. Emotional availability: conceptualization and research findings. Am J Orthopsychiatry. 2000 Jan;70(1):104-14. doi: 10.1037/h0087711. PMID 10702855
- [Background] Bowlby J. Attachment and loss: retrospect and prospect. Am J Orthopsychiatry. 1982 Oct;52(4):664-678. doi: 10.1111/j.1939-0025.1982.tb01456.x. No abstract available. PMID 7148988
- [Background] Bowlby, J. A Secure Base. doi:Basic Books (1988).
- [Background] Biringen Z, Robinson JL, Emde RN. Appendix A: the emotional availability scales (2nd ed.; an abridged infancy/Early Childhood version). Attach Hum Dev. 2000 Sep;2(2):251-70. doi: 10.1080/14616730050085617. No abstract available. PMID 11707915
- [Background] Bornstein MH, Gini M, Putnick DL, Haynes OM, Painter KM, Suwalsky JTD. Short-Term Reliability and Continuity of Emotional Availability in Mother-Child Dyads Across Contexts of Observation. Infancy. 2006 Jul;10(1):1-16. doi: 10.1207/s15327078in1001_1. Epub 2006 Jul 1. PMID 33412671
- [Background] Buss C, Lord C, Wadiwalla M, Hellhammer DH, Lupien SJ, Meaney MJ, Pruessner JC. Maternal care modulates the relationship between prenatal risk and hippocampal volume in women but not in men. J Neurosci. 2007 Mar 7;27(10):2592-5. doi: 10.1523/JNEUROSCI.3252-06.2007. PMID 17344396
- [Background] Barnat SB, Klein PJ, Meltzoff AN. Deferred Imitation Across Changes in Context and Object: Memory and Generalization in 14-Month-Old Infants. Infant Behav Dev. 1996 Apr 1;19(2):241-251. doi: 10.1016/S0163-6383(96)90023-5. PMID 25147417
- [Background] Olds D, Henderson CR Jr, Kitzman H, Cole R. Effects of prenatal and infancy nurse home visitation on surveillance of child maltreatment. Pediatrics. 1995 Mar;95(3):365-72. PMID 7862474
- [Background] Olds DL, Kitzman H, Cole R, Robinson J, Sidora K, Luckey DW, Henderson CR Jr, Hanks C, Bondy J, Holmberg J. Effects of nurse home-visiting on maternal life course and child development: age 6 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1550-9. doi: 10.1542/peds.2004-0962. PMID 15574614